CLINICAL TRIAL: NCT07148440
Title: Frequency and Types of Acid-Base Disorders in Intensive Care Unit Patients
Brief Title: Acid Base Disorders in ICU in Minia University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sohair Adeeb, assistant professor, Minia University
Other Study IDs: Acid base disorders in ICU
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Septicemia
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data extracted from records of patients in the ICU regarding type and frequency of acid base disturbance that led to their admission to the ICU and correlation with 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission with documented acid base disturbance

Exclusion Criteria:

* incomplete records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all icu patients with acid base abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-08-23 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Types of acid- base disorders in ICU patients | from January 2021 to December 2024

SECONDARY OUTCOMES:
28 day mortality | from January 2021 to December 2024

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achanti A, Szerlip HM. Acid-Base Disorders in the Critically Ill Patient. Clin J Am Soc Nephrol. 2023 Jan 1;18(1):102-112. doi: 10.2215/CJN.04500422. Epub 2022 Aug 23. PMID 35998977